CLINICAL TRIAL: NCT03625427
Title: Effects of Palmitoleic Acid on Circulating C-reactive Protein Levels in Humans
Brief Title: Effect of Palmitoleic Acid on C-reactive Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Organic Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-2316
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Chronic Inflammation; Overweight
Keywords: palmitoleic acid; monounsaturated fatty acid; chronic inflammation
MeSH Terms: conditions — Overweight | interventions — Olive Oil; palmitoleic acid

STUDY DESIGN:
Intervention Model Description: 12-week randomized, double blinded study in volunteers consuming either the test agent, 500 mg or 1,000 mg POA per day, or an olive oil containing fatty acid (placebo). There are three arms to study and 41 individuals per arm, thus, a total of 123 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Administration of the POA supplements and placebo (olive oil capsules) will be via a simple randomized double-blinded allocation. The study sponsor will provide the Principal Investigator with bags, or boxes, of single serve packets containing two capsules for each daily dose per participant in accordance with the proper dosage for each of the three arms of the study. The study sponsor will hold the code for the subjects and will randomize the capsules. No site personnel will have access to the randomization allocation; only the study sponsor will have the code. The identity of the capsules will be revealed once all analyses are complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo is olive oil, stripped of polyphenols, 70% oleic acid, and will be administered at two 1 gram capsules per day for twelve weeks. The doses will be administered in single serve packets containing two capsules for each daily dose to be taken at breakfast.
  Interventions: Dietary Supplement: Placebo
- Palmitoleic acid, 500 mg (Dose 1) (Experimental): POA Dose 1 is a 1 gram capsule containing 500 mg POA and one placebo capsule containing 500 mg olive oil per day for twelve weeks. The doses will be administered in single serve packets containing two capsules for each daily dose to be taken at breakfast.
  Interventions: Dietary Supplement: Palmitoleic acid, 500 mg (Dose 1)
- Palmitoleic acid, 1,000 mg (Dose 2) (Experimental): POA Dose 2 is two, 1 gram capsules containing 500 mg POA, totaling 1,000 mg POA per day for twelve weeks.The doses will be administered in single serve packets containing two capsules for each daily dose to be taken at breakfast.
  Interventions: Dietary Supplement: Palmitoleic acid, 1,000 mg (Dose 2)

INTERVENTIONS:
Dietary Supplement: Placebo — The placebo is olive oil, stripped of polyphenols, 70% oleic acid, administered as two 1-gram capsules per day. Packaged as single-serve packets containing 2 capsules for each daily dose.
  Other Names: Olive oil
  Arms: Placebo
Dietary Supplement: Palmitoleic acid, 500 mg (Dose 1) — Palmitoleic acid (POA) 1 gram capsules containing 500 mg POA
  Other Names: POA
  Arms: Palmitoleic acid, 500 mg (Dose 1)
Dietary Supplement: Palmitoleic acid, 1,000 mg (Dose 2) — Palmitoleic acid (POA) taken as two 1 gram capsules each containing 500 mg POA
  Other Names: POA
  Arms: Palmitoleic acid, 1,000 mg (Dose 2)

SUMMARY:
This clinical trial will test the effects of an n-7 monounsaturated fatty acid known as palmitoleic acid (POA) on a chronic inflammation marker in overweight subjects. The study will enroll male and female subjects from healthy populations with high levels of the inflammatory marker c-reactive protein (CRP). Investigators will then determine over time if palmitoleic acid supplementation can lower circulating levels of c-reactive protein. Investigators will administer palmitoleic acid at two doses in addition to a placebo and conduct a double-blind parallel arm study. Circulating CRP will be the primary endpoint and secondary endpoints are Interleukin 6 (IL-6), Tumor necrosis factor (TNF) alpha, ghrelin, peptide tyrosine tyrosine (peptide YY), cardio lipid markers, glucose, insulin, leptin, adiponectin, and red blood cell (RBC) and serum fatty acids.

DETAILED DESCRIPTION:
Palmitoleic acid (POA) is a monounsaturated fatty acid that has recently been shown to function as a lipokine and is present in the human diet and in blood serum. While there is emerging evidence that POA can positively impact beta cell proliferation, reduce lipogenesis, support endothelial function, and suppress cytokine production, POA remains to be poorly studied for its beneficial anti-inflammatory potential. The latest studies suggest that POA could attenuate inflammation in metabolically active tissues. Therefore, the objective of this study is to determine if administration of POA in 2 varying doses to overweight participants with biomarkers of chronic inflammation will lower circulating c-reactive protein (CRP) and cytokine levels, as well as improve metabolism by lowering levels of circulating leptin and raising expression of adiponectin. The rationale for focusing on overweight individuals is that they routinely have elevated c-reactive protein levels and are highly prone to have chronic inflammation.

Investigators propose a 12-week randomized, double blinded study to assess changes in select inflammatory markers, ghrelin, peptide YY, cardiovascular lipids, fatty acid levels, and glucose sensitivity markers in volunteers consuming either the test agent, 500 mg or 1,000 mg POA per day, or an olive oil containing fatty acid (placebo). There are three arms to study and 41 individuals per arm, thus, a total of 123 subjects. Approximately 30% loss of subjects is expected. Administration of the POA supplements and placebo (olive oil capsules) will be double blinded. The study sponsor will hold the code for the subjects and will randomize the capsules. Only the study sponsor will have the code. The identity of the capsules will be revealed after the completion of the study. Subjects will bring back their bottles at each of the concurrent visits and the end of the study to assess compliance and to account for any missed doses of POA. The rationale for selecting olive oil as a placebo is that olive oil is routinely consumed by the public. Additionally, oleic acid (the active ingredient of olive oil) is the most prevalent fatty acid in human circulation, and olive oil is a routine placebo for fatty acid intervention studies. The olive oil will not be extra virgin olive oil that has several bioactive components. POA is virtually tasteless, thus participants should not be able to self-identify their regimen of either placebo or active test agent. The rationale for the experimental dose follows what is commercially available in POA products, which average 700 mg per day and generally range from 450 - 1000 mg per day regimens. The rationale for the 12-week time frame is to ensure uptake of POA into the target cells.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be free-living, middle-aged to older men and women between ages 18-80 years with BMIs between 20.0-40.0, and CRP greater than or equal to 2.0 mg/L
2. Generally healthy adults
3. Understand protocol and comply to take supplements during the trial
4. Ability to understand English
5. Be able to report to clinical research center, fasting, at least 3 times
6. Women who are of childbearing potential should be on birth control (one method is acceptable)

Exclusion Criteria:

1. BMI higher than 40.0
2. Taking anti-hyperlipidemia medications (including statins)
3. Taking anti-diabetic medications
4. Auto-immune disease
5. Documented cognitive impairment
6. Unable to draw blood from veins
7. Alcohol or other drug dependency
8. Are currently breastfeeding, or pregnant, or plan to become pregnant
9. Have experienced a significant weight change of 10%, or more, of body weight in previous 3 months
10. If on hormone therapy, no change during study
11. Chronic use of NSAIDs
12. Decreased QOL due to pathology, such as cancer, genetic diseases, Rx side effects, or injury
13. Taking fish oil, within 8 weeks of enrollment
14. Taking Seabuckthorn supplements
15. Taking sterols or fat blockers
16. Fish allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Mean c-reactive protein circulating level | Week 12
  Fasting blood draws will be used to evaluate circulating CRP level by high-sensitivity c-reactive protein laboratory blood analysis.

SECONDARY OUTCOMES:
Mean circulating cytokine IL-6 level | Week 12
  Fasting blood draws will be used to evaluate circulating cytokine IL-6 level by ELISA (enzyme-linked immunosorbent assay).
Mean circulating cytokine TNF alpha level | Week 12
  Fasting blood draws will be used to evaluate circulating cytokine TNF alpha level by ELISA (enzyme-linked immunosorbent assay).
Mean circulating ghrelin level | Week 12
  Fasting blood draws will be used to evaluate circulating ghrelin level by ELISA (enzyme-linked immunosorbent assay).
Mean circulating peptide YY level | Week 12
  Fasting blood draws will be used to evaluate circulating peptide YY level by ELISA (enzyme-linked immunosorbent assay).
Mean circulating leptin level | Week 12
  Fasting blood draws will be used to evaluate circulating leptin level by ELISA (enzyme-linked immunosorbent assay).
Mean circulating adiponectin level | Week 12
  Fasting blood draws will be used to evaluate circulating adiponectin level by ELISA (enzyme-linked immunosorbent assay).
Mean glucose/insulin ratio level | Week 12
  Fasting blood draws will be used to evaluate glucose/insulin ratio level.
Mean HbA1c level | Week 12
  Fasting blood draws will be used to evaluate HbA1c level.

CONTACTS AND LOCATIONS:
Overall Officials: Saame R Shaikh, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication.
Access Criteria: A Data Use Agreement (DUA) specifying the uses of such data to be shared must be in place before any data is shared. The requestor should contact the Principal Investigator for further instruction.

REFERENCES:
- [Background] Frigolet ME, Gutierrez-Aguilar R. The Role of the Novel Lipokine Palmitoleic Acid in Health and Disease. Adv Nutr. 2017 Jan 17;8(1):173S-181S. doi: 10.3945/an.115.011130. Print 2017 Jan. PMID 28096141
- [Background] Yadav A, Kataria MA, Saini V, Yadav A. Role of leptin and adiponectin in insulin resistance. Clin Chim Acta. 2013 Feb 18;417:80-4. doi: 10.1016/j.cca.2012.12.007. Epub 2012 Dec 22. PMID 23266767
- [Background] Schirmer M, Smeekens SP, Vlamakis H, Jaeger M, Oosting M, Franzosa EA, Ter Horst R, Jansen T, Jacobs L, Bonder MJ, Kurilshikov A, Fu J, Joosten LAB, Zhernakova A, Huttenhower C, Wijmenga C, Netea MG, Xavier RJ. Linking the Human Gut Microbiome to Inflammatory Cytokine Production Capacity. Cell. 2016 Nov 3;167(4):1125-1136.e8. doi: 10.1016/j.cell.2016.10.020. PMID 27814509
- [Background] de Souza CO, Vannice GK, Rosa Neto JC, Calder PC. Is Palmitoleic Acid a Plausible Nonpharmacological Strategy to Prevent or Control Chronic Metabolic and Inflammatory Disorders? Mol Nutr Food Res. 2018 Jan;62(1). doi: 10.1002/mnfr.201700504. Epub 2017 Dec 11. PMID 28980402
- [Result] Bernstein AM, Roizen MF, Martinez L. WITHDRWAN: Purified palmitoleic acid for the reduction of high-sensitivity C-reactive protein and serum lipids: a double-blinded, randomized, placebo controlled study. J Clin Lipidol. 2014 Nov-Dec;8(6):612-617. doi: 10.1016/j.jacl.2014.08.001. Epub 2014 Aug 19. PMID 25499944 (Retraction: PMID 34144766 J Clin Lipidol. 2021 May-Jun;15(3):522)